CLINICAL TRIAL: NCT03612232
Title: A Multicenter, Open-label, Phase II Study to Evaluate the Efficacy and Safety of Cabozantinib in Advanced (Unresectable or Metastatic) Adrenocortical Carcinoma
Brief Title: Cabozantinib in Advanced Adrenocortical Carcinoma
Acronym: CaboACC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboACC
Record Dates: First submitted 2018-07-12; First posted 2018-08-02 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-12

CONDITIONS: Adrenocortical Carcinoma
Keywords: adrenal cancer; adrenal cortex neoplasm; adrenal cortical carcinoma; cabozantinib; c-MET
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms; Adrenal Cortex Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cabozantinib (Experimental): oral cabozantinib as tablets continuously (60 mg single dose, tablets)
  Interventions: Drug: Cabozantinib-s-malate

INTERVENTIONS:
Drug: Cabozantinib-s-malate — oral cabozantinib-S-malate 60 mg as a daily single oral dose continuously

SUMMARY:
Adrenocortical carcinoma is an orphan malignant disease that has a dismal prognosis in advanced stages. Mitotane is the only approved treatment but is limited by severe toxicity. Efficacy of mitotane is unsatisfactory with an objective response rate of ≈20% in monotherapy in selected patients (Megerle et al., JCEM 2018). Cytotoxic chemotherapy with etoposide, doxorubin and cisplatin (EDP) or streptozotocin (Sz) in addition to mitotane (Fassnacht et al., N Engl J Med 2012) succeeded in a progression-free survival of 5.6 months and 2.2 months, respectively in patients with advanced ACC. Objective response rates were 23 and 9%. EDP plus mitotane is therefore considered as standard treatment of ACC. Results by Phan et al. (Cancer Research 2015) demonstrated expression of c-MET and its ligand HGF in ACC and provide a rationale to therapeutically target c-MET in ACC. In a case series of 16 patients with advanced ACC refractory to mitotane (with the exception of one case) and 3 (median, range 0-8)further lines of therapy, single agent treatment with cabozantinib off label resulted in three partial responses and five additional cases of disease stabilization for four months or longer (Kroiss et al., J Clin Endocrinol Metab 2020).

ELIGIBILITY:
Inclusion criteria:

* Histological confirmation of ACC based on either:

  i) Weiss Score of ≥ 3 in patients who had earlier surgical resection (Lin-Weiss-Bisceglia system will be used for oncocytic ACC) OR ii) biopsy results compatible with ACC in the context of clinical setting highly suggestive of ACC (adrenal mass > 4 cm invading surrounding organs or associated with distant metastases).
* Locally advanced or metastatic disease not amenable to surgery with curative intent with measurable disease per RECIST 1.1 37 as determined by the investigator based on an assessment of all known disease sites by computerized tomography (CT) scan or magnetic resonance imaging (MRI) of chest/abdomen/pelvis within 28 days before the first dose of cabozantinib
* Received prior treatment with mitotane and platinum containing chemotherapy. Patients in whom mitotane and/or platinum containing chemotherapy is contraindicated or who refused treatment with mitotane and/or platinum containing chemotherapy are eligible for the study.
* Documented progressive disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Recovery to baseline or ≤ Grade 1 CTCAE v.5.0 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy
* Life expectancy of at least 3 months
* Adequate organ and bone marrow function and laboratory values as follows within 14 days prior to the first dose of cabozantinib:

  1. Absolute neutrophil count (ANC) ≥ 1500/μL without colony stimulating factor support, white blood cell count ≥ 2500/μL.
  2. Platelets ≥ 100,000/μL without transfusion
  3. Hemoglobin ≥ 9 g/dL
  4. Bilirubin ≤ 1.5 × the upper limit of normal (ULN). For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL
  5. Serum albumin ≥ 2.8 g/dl
  6. (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN
  7. Serum creatinine ≤ 2.0 × ULN or creatinine clearance (CrCl) ≥ 30 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

     Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72). Female:

     Multiply above result by 0.85
  8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). In case of liver metastases ALT and AST ≤ 5.0 x ULN are acceptable. ALP ≤ 5 x ULN with documented bone metastases.
  9. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg), or 24-h urine protein ≤ 1 g
* Capable of understanding and complying with the protocol requirements.
* Women of childbearing potential* must have a negative pregnancy test at screening.

Additional pregnancy testing will be performed in WOCBP at monthly intervals. Patients of reproductive potential (men and women) must agree to use highly effective methods of contraception during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. - Able to give written informed consent

Exclusion criteria:

* Received cytotoxic chemotherapy, or targeted therapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies), or other investigational agent within 14 days before study treatment.
* Treatment with mitotane <28 days prior study inclusion OR mitotane serum/plasma concentration documented of ≥2 mg/L at screening. Up to 5 mg/L are acceptable with Sponsor approval.
* Prior treatment with cabozantinib or other cMET inhibitors
* Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment (eg, I-131 or Y-90) within 6 weeks before first dose of study treatment.

Subject is excluded if there are any clinically relevant ongoing complications from prior radiation therapy.

- Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis).

Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.

Corticosteroid replacement treatment is allowed with dose at the discretion of the investigator.

* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* The use of strong CYP3A4 inhibitors (with the exception of ketoconazole).
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias. ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment. b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction. ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels. In subjects with liver metastases and lesions invading the intrahepatic vasculature, including portal vein, hepatic vein, and hepatic artery, are eligible
* Other clinically significant disorders that would preclude safe study participation.

  1. Serious non-healing wound/ulcer/bone fracture.
  2. Uncompensated/symptomatic hypothyroidism.
  3. Severe and uncontrolled Cushing's syndrome despite medical management (e.g. systolic blood pressure >160 mmHg, hyperglycemia with fasting glucose >300 mg/dL)
  4. Moderate to severe hepatic impairment (Child-Pugh B or C).
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) or dental surgery/invasive dental procedures within 28 days before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment [add reference for Fridericia formula].
* Pregnant or lactating females
* Inability to swallow tablets.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 2 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality which, in the judgment of the investigator, would have made the patient inappropriate for entry into this study
* Any other severe acute or chronic medical or psychiatric condition or laboratory ab normality which, in the judgment of the investigator, would have made the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival at 4 months | 4 months

SECONDARY OUTCOMES:
Objective Response Rates (ORR) | 12 months
Duration of response (DR) | 12 months
progression-free survival | 12 months
overall survival | 12 months
best percentage change in size of target lesions | 12 months
treatment emergent adverse events (CTC-AE 4.03) | 12 months
quality of life by EORTC QLQ-C30 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kroiss, MD, PhD, Study Director — Wuerzburg University Hospital
Locations (2):
- Germany (2):
  - University Hospital Munich, Department of Internal Medicine IV, München
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan LM, Fuentes-Mattei E, Wu W, Velazquez-Torres G, Sircar K, Wood CG, Hai T, Jimenez C, Cote GJ, Ozsari L, Hofmann MC, Zheng S, Verhaak R, Pagliaro L, Cortez MA, Lee MH, Yeung SC, Habra MA. Hepatocyte Growth Factor/cMET Pathway Activation Enhances Cancer Hallmarks in Adrenocortical Carcinoma. Cancer Res. 2015 Oct 1;75(19):4131-42. doi: 10.1158/0008-5472.CAN-14-3707. Epub 2015 Aug 17. PMID 26282167
- [Background] Kroiss M, Megerle F, Kurlbaum M, Zimmermann S, Wendler J, Jimenez C, Lapa C, Quinkler M, Scherf-Clavel O, Habra MA, Fassnacht M. Objective Response and Prolonged Disease Control of Advanced Adrenocortical Carcinoma with Cabozantinib. J Clin Endocrinol Metab. 2020 May 1;105(5):1461-8. doi: 10.1210/clinem/dgz318. PMID 31900481
- See also: Wuerzburg University Hospital — http://ukw.de